CLINICAL TRIAL: NCT02155543
Title: A Safety, Tolerability, and Pharmacokinetics (PK) Study of AGN-223575 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 223575-001
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Cohort 1: AGN-223575 Form A/Vehicle (Experimental): One drop of AGN-223575 Formulation A in the study eye and one drop of AGN-223575 vehicle in the other eye on day 1, followed by one drop of AGN-223575 Formulation A twice daily in the study eye and 1 drop of AGN-223575 vehicle in the other eye twice daily for 6 days.
  Interventions: Drug: AGN-223575 Formulation A; Drug: AGN-223575 Vehicle
- Cohort 2: AGN-223575 Formulation A BID (Experimental): One drop of AGN-223575 Formulation A in both eyes on day 1, followed by one drop of AGN-223575 Formulation A twice daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation A in both eyes on day 15.
  Interventions: Drug: AGN-223575 Formulation A
- Cohort 3: AGN-223575 Formulation B BID (Experimental): One drop of AGN-223575 Formulation B in both eyes on day 1, followed by one drop of AGN-223575 Formulation B twice daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation B in both eyes on day 15.
  Interventions: Drug: AGN-223575 Formulation B
- Cohort 4: AGN-223575 Formulation C BID (Experimental): One drop of AGN-223575 Formulation C in both eyes on day 1, followed by one drop of AGN-223575 Formulation C twice daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation C in both eyes on day 15.
  Interventions: Drug: AGN-223575 Formulation C
- AGN-223575 Vehicle BID (Placebo Comparator): One drop of AGN-223575 vehicle in both eyes on day 1, followed by one drop of AGN-223575 vehicle twice daily in both eyes for 13 days, and a single drop of AGN-223575 vehicle in both eyes on day 15.
  Interventions: Drug: AGN-223575 Vehicle
- Cohort 5: AGN-223575 Formulation C TID (Experimental): One drop of AGN-223575 Formulation C in both eyes on day 1, followed by one drop of AGN-223575 Formulation C three times daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation C in both eyes on day 15.
  Interventions: Drug: AGN-223575 Formulation C
- AGN-223575 Vehicle TID (Placebo Comparator): One drop of AGN-223575 vehicle in both eyes on day 1, followed by one drop of AGN-223575 vehicle three times daily in both eyes for 13 days, and a single drop of AGN-223575 vehicle in both eyes on day 15.
  Interventions: Drug: AGN-223575 Vehicle

INTERVENTIONS:
Drug: AGN-223575 Formulation A — One drop of AGN-223575 Formulation A administered in the study eye(s) per protocol.
  Arms: Cohort 1: AGN-223575 Form A/Vehicle; Cohort 2: AGN-223575 Formulation A BID
Drug: AGN-223575 Formulation B — One drop of AGN-223575 Formulation B in both eyes on day 1, followed by one drop of AGN-223575 Formulation B twice daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation B in both eyes on day 15.
  Arms: Cohort 3: AGN-223575 Formulation B BID
Drug: AGN-223575 Formulation C — One drop of AGN-223575 Formulation C in both eyes on day 1, followed by one drop of AGN-223575 Formulation C twice daily in both eyes for 13 days, and a single drop of AGN-223575 Formulation C in both eyes on day 15.
  Arms: Cohort 4: AGN-223575 Formulation C BID; Cohort 5: AGN-223575 Formulation C TID
Drug: AGN-223575 Vehicle — One drop of AGN-223575 vehicle administered in the study eye(s) per protocol.
  Arms: AGN-223575 Vehicle BID; AGN-223575 Vehicle TID; Cohort 1: AGN-223575 Form A/Vehicle

SUMMARY:
This study will evaluate the safety, tolerability, and pharmacokinetics (PK) of AGN-223575 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Weight at least 110 lbs

Exclusion Criteria:

* Use of contact lenses within 14 days, or planned use during the study
* Use of any ocular eye medications within 30 days, or anticipated use during the study
* Anticipated use of any artificial tears product during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Newport Beach, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 5: AGN-223575 Formulation C TID | Cohort 4: AGN-223575 Formulation C BID | Cohort 3: AGN-223575 Formulation B BID | Cohort 2: AGN-223575 Formulation A BID | Cohort 1: AGN-223575 Form A/Vehicle | AGN-223575 Vehicle TID | AGN-223575 Vehicle BID
Started | 9 | 9 | 9 | 9 | 3 | 3 | 9
Completed | 9 | 9 | 9 | 9 | 3 | 3 | 9
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 5: AGN-223575 Formulation C TID | Cohort 4: AGN-223575 Formulation C BID | Cohort 3: AGN-223575 Formulation B BID | Cohort 2: AGN-223575 Formulation A BID | Cohort 1: AGN-223575 Form A/Vehicle | AGN-223575 Vehicle TID | AGN-223575 Vehicle BID | Total
Number analyzed (Participants) | 9 | 9 | 9 | 9 | 3 | 3 | 9 | 51
Age, Customized [Number; unit: Participants]
  <45 years | 7 | 8 | 9 | 9 | 3 | 3 | 9 | 48
  Between 45 and 65 years | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 3 | 6 | 5 | 1 | 2 | 5 | 31
  Male | 0 | 6 | 3 | 4 | 2 | 1 | 4 | 20

OUTCOME MEASURES:

1. Primary Outcome: Maximal Plasma Concentration (Cmax) of AGN-223575
Description: Concentrations of AGN-223575 were measured in the plasma (the liquid component of the blood in which the blood cells are suspended) in samples collected up to 24 hours post-dose. The Cmax is reported.
Time Frame: Day 15
Population: Pharmacokinetic Population: AGN-223575-treated subjects in cohorts with pharmacokinetic samples (i.e., Cohorts 2 to 5)
Measure: Mean (Standard Deviation); unit: Nanograms/Milliliters (ng/mL)
Arm/Group | Cohort 5: AGN-223575 Formulation C TID | Cohort 4: AGN-223575 Formulation C BID | Cohort 3: AGN-223575 Formulation B BID | Cohort 2: AGN-223575 Formulation A BID
Number analyzed (Participants) | 9 | 9 | 9 | 9
Nanograms/Milliliters (ng/mL) | 0.186 (0.095) | 0.128 (0.060) | 0.114 (0.085) | NA (NA) — Data were below the limit of quantitation (< 0.02 ng/mL)

ADVERSE EVENTS:
Description: The Safety Population included all subjects who received study drug (or vehicle) and was used to assess adverse events and serious adverse events.
Arm/Group | Cohort 5: AGN-223575 Formulation C TID | Cohort 4: AGN-223575 Formulation C BID | Cohort 3: AGN-223575 Formulation B BID | Cohort 2: AGN-223575 Formulation A BID | AGN-223575 Vehicle TID | AGN-223575 Vehicle BID | Cohort 1: AGN-223575 Form A/Vehicle
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/9 | 0/9 | 0/9 | 0/3 | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 2/9 | 1/9 | 2/9 | 0/9 | 0/3 | 1/9 | 0/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 5: AGN-223575 Formulation C TID (N=9) | Cohort 4: AGN-223575 Formulation C BID (N=9) | Cohort 3: AGN-223575 Formulation B BID (N=9) | Cohort 2: AGN-223575 Formulation A BID (N=9) | AGN-223575 Vehicle TID (N=3) | AGN-223575 Vehicle BID (N=9) | Cohort 1: AGN-223575 Form A/Vehicle (N=3)
Punctate Keratitis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0
Eye Discharge (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Intraocular Pressure Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Instillation Site Pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.